CLINICAL TRIAL: NCT05936398
Title: Influence of Respiratory Muscle Training on Objective and Subjective Training Load Measures in Triathletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Sport - National Research Institute, Poland (Other)
Responsible Party: Principal Investigator, Tomasz Kowalski, Specialist, Institute of Sport - National Research Institute, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TK02/2023
Record Dates: First submitted 2023-06-23; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Athletic Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voluntary Isocapnic Hyperpnoea (VIH) (Active Comparator): Group performing respiratory muscle training with Voluntary Isocapnic Hyperpnoea (VIH) method.
  Interventions: Behavioral: Respiratory Muscle Training - VIH
- Inspiratory Pressure Threshold Loading (IPTL) (Active Comparator): Group performing respiratory muscle training with Inspiratory Pressure Threshold Loading (IPTL) method.
  Interventions: Behavioral: Respiratory Muscle Training - ITPL

INTERVENTIONS:
Behavioral: Respiratory Muscle Training - VIH — The VIH group will train every second day with gradual progression based on session length and breathing frequency. Participants will begin with 3 minutes of exercise with a frequency of 20 breaths·min-1 during the first session and add no more than 1 minute or 2 breaths·min-1 with each consecutive session.
  Arms: Voluntary Isocapnic Hyperpnoea (VIH)
Behavioral: Respiratory Muscle Training - ITPL — The IPTL group will train 5 days a week, twice a day, with at least 6 hours break between sessions. The session will consist of 30 dynamic inspiratory maneuvers with progressive overload based on gradually increased resistance. The VIH group will train every second day with gradual progression based on session length and breathing frequency. Participants will begin with 3 minutes of exercise with a frequency of 20 breaths·min-1 during the first session and add no more than 1 minute or 2 breaths·min-1 with each consecutive session.
  Arms: Inspiratory Pressure Threshold Loading (IPTL)

SUMMARY:
Two groups of healthy, highly trained triathletes trained respiratory muscles with one of the two methods: voluntary isocapnic hyperpnoea (VIH) or inspiratory pressure threshold loading (IPTL). The main purpose of this study was to accurately and thoroughly assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods.

Informed written consent was obtained from the all study participants. All procedures were carried out in accordance with the Declaration of Helsinki.

DETAILED DESCRIPTION:
The study was conducted as a randomized controlled trial with two parallel groups. Whereas participants and data collectors were aware of the allocated training method, the data analysts and laboratory technicians performing biochemistry assays were kept blinded to the allocation. The participants were assigned at random to either VIH or IPTL training group to perform RMT with progressive overload for 6 weeks.

Three training sessions (week 1, 4, 6) were monitor to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods.

Blood samples used for acid-base balance (pH), partial pressure of oxygen (pO2), partial pressure for carbon dioxide (pCO2), partial pressure for bicarbonate ion (HCO3-), and blood lactate (bLa) were collected immediately after cessation of the exercise and MPQ was presented 1' after cessation of the exercise. Blood samples for cortisol (C) and testosterone (T) were collected 5' after cessation of the exercise. The second S-Index Test was performed between minute 5 and minute 7 after cessation of the exercise. RPE was assessed 10' after cessation of the exercise. The participants again answered MPQ after 24h and 48h after the monitored RMT sessions.

Informed written consent was obtained from the all study participants. All procedures were carried out in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* valid medical certificate to compete sports professionally,
* lack of ongoing medication intake,
* lack of any medical condition,
* lack of previous experience with RMT,
* lack of previous experience with RMT,
* performance caliber corresponding to at HighlyTrained/Elite (Participant Classification Framework, McKay 2022),
* at least 6 years of triathlon training,
* average training volume over 12 hours per week during last 6 weeks.

Exclusion Criteria:

* any ongoing medication intake or medical condition.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in measured blood indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (pH) | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in pre- and post- RMT session in pH.
Changes in measured blood indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (pO2). | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in pre- and post- RMT session in pO2.
Changes in measured blood indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (pCO2). | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in pre- and post- RMT session in pCO2.
Changes in measured blood indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (CHO3). | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in pre- and post- RMT session in CHO3. CHO3.
Changes in measured blood indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (lactate). | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in pre- and post- RMT session in blood lactate levels.
Changes in measured blood indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (testosterone). | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in pre- and post- RMT session in testosterone.
Changes in measured blood indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (cortisol). | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in pre- and post- RMT session in cortisol.
Changes in cardiac indices to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods. | Week 1, 4 and 6 after monitored RMT sessions.
  Differences in HR indices between methods, increase of HR and decrease of HR after the cessation on the exercise.
Collecting subjective measures to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (RPE) | Week 1, 4 and 6 after monitored RMT sessions.
  Collecting perceived exertion numbers (Rate of Perceived Exertion - RPE)
Collecting subjective measures to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods (MPQ). | Week 1, 4 and 6 after monitored RMT sessions.
  Collecting McGill Pain Questionnaire immediately post-session (MPQ scale).
Collecting local blood oxygenation during RMT to assess the potential extra load that RMT puts on athletes and determine if there are significant differences in RMT-induced load between the investigated training methods. | Week 1, 4 and 6 after monitored RMT sessions.
  Measuring SMO2 before, during and after RMT sessions to assess induced changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sport - National Research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No